CLINICAL TRIAL: NCT03457688
Title: Double-blind, Randomized Placebo-controlled, Multi-center Trial Investigating the Effect of Prebiotic Inulin-type Fructans on Infectious Incidence in Children Aged 3 to 6 Years
Brief Title: Effect of Prebiotic Fructans to Reduce Number of Febrile Infections in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo-Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16002n_
Record Dates: First submitted 2018-02-21; First posted 2018-03-07 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Infectious Disease; Children, Only; Diet Modification
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prebiotic inulin-type fructans (Active Comparator)
  Interventions: Dietary Supplement: prebiotic inulin-type fructans
- placebo maltodextrin (Placebo Comparator)
  Interventions: Dietary Supplement: placebo maltodextrin

INTERVENTIONS:
Dietary Supplement: prebiotic inulin-type fructans
  Arms: prebiotic inulin-type fructans
Dietary Supplement: placebo maltodextrin
  Arms: placebo maltodextrin

SUMMARY:
The study aims to confirm the effectiveness of chicory-derived prebiotic inulin-type fructans on the reduction of the number of febrile infections diagnosed by the paediatrician in children.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy at the time of pre-examination
* Subject is aged 3-6 years at the time of pre-examination
* Subject attends a kindergarten at the time of pre-examination

Exclusion Criteria:

* Suffering from current infection or has suffered from infection in previous 7 days
* Intake of antibiotics and/or laxatives in the previous 14 days prior to start of the intervention
* children with known gastrointestinal disease or malformation
* children with congenital or acquired immunodeficiency
* children with food intolerance, food allergy
* children that regularly consume (more than 3 times per week) probiotic products or a food supplement containing prebiotics
* children involved in any clinical or food study within the preceding 6 months

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 850 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Number of febrile infectious episodes diagnosed by paediatrician | 6 months period

SECONDARY OUTCOMES:
Number of any infectious episodes diagnosed by paediatrician | 6 months period
Number of episodes with symptoms of illnesses indicating a viral or bacterial infection | 6 months period
Duration of febrile infectious episodes diagnosed by the paediatrician | 6 months period
Duration of any infectious episode | 6 months period
Duration of episodes with symptoms of illnesses indicating a viral or bacterial infection | 6 months period
Days of absence from day-care of the child due to infectious episodes and/or symptoms of dysbiosis (diarrhoea) following antibiotic treatment | 6 months period
Number of paediatrician´s consultations due to infectious disease and/ or symptoms of dysbiosis (diarrhoea) following antibiotic treatment | 6 months period
Hospitalization days due to infectious disease and/or symptoms of dysbiosis | 6 months period
Number of days (parents questionnaire and diary) of caretaker´s absenteeism from work due to infectious episodes and/or symptoms of dysbiosis of the child | 6 months period
Number of episodes on antibiotic treatment | 6 months period
Number of days on antibiotic treatment | 6 months period
Number of episodes of medication use (including prescribed/ non-prescribed medication and antibiotics/ non-antibiotics) | 6 months period
Number of days of medication use (including prescribed/ non-prescribed medication and antibiotics/ non-antibiotics) | 6 months period
Quality of life reported by the parents according to standardized questionnaire | 6 months period
  Parent Diary (scale: no, minor, moderate, significant changes, Not known)
Analysis of stool samples in a subset of children: microbiota changes | 6 months period

OTHER OUTCOMES:
Incidence of gastrointestinal discomfort | 6 months period
  Main Parameters of safety
Body Weight | 6 months period
  Main Parameters of safety
Body Height | 6 months period
  Main Parameters of safety
Side effects (Questionnaire) | 6 months period
  Main Parameters of safety

CONTACTS AND LOCATIONS:
Overall Officials: Tamás Decsi, Prof., Principal Investigator — Department of Paediatrics, University of Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lohner S, Kullenberg D, Antes G, Decsi T, Meerpohl JJ. Prebiotics in healthy infants and children for prevention of acute infectious diseases: a systematic review and meta-analysis. Nutr Rev. 2014 Aug;72(8):523-31. doi: 10.1111/nure.12117. Epub 2014 Jun 5. PMID 24903007